CLINICAL TRIAL: NCT06139692
Title: Comparison of Perioperative Conscious Sedation During Endovascular Thrombectomy in Acute Ischemic Stroke (PEACE) A Randomised Multicentre Trial
Brief Title: Comparison of Perioperative Conscious Sedation During Endovascular Thrombectomy in Acute Ischemic Stroke
Acronym: PEACE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Xinfeng Liu, Professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEACE
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the dexmedetomidine group (Experimental): In the experimental group, dexmedetomidine is used for intraoperative sedation. Dexmedetomidine is prepared as an 8μg/ml intravenous infusion. It begins with an initial loading dose of 1μg/kg, administered over a period exceeding 10 minutes.If dexmedetomidine fails to achieve a satisfactory level of sedation during surgery, physicians may opt for rescue sedation with propofol or consider transferring the patient to general anesthesia. Propofol (20ml 0.2g) starts with a loading dose of 0.3mg/(kg*h) and a maintenance dose of 0.3-4mg/(kg*h). The infusion rate can be adjusted based on the sedation effect to achieve the appropriate level of sedation during EVT.
  Interventions: Drug: Dexmedetomidine
- the midazolam group (Active Comparator): In the control group, midazolam is used for intraoperative sedation. Midazolam is prepared as a 1mg/ml intravenous infusion. It starts with an initial intravenous push of 0.05mg/kg, followed by a maintenance dose of 0.04-0.2mg/kg administered intravenously via an infusion pump. If midazolam fails to achieve a satisfactory level of sedation during surgery, physicians may opt for rescue sedation with propofol or consider transferring the patient to general anesthesia. Propofol (20ml 0.2g) starts with a loading dose of 0.3mg/(kg*h) and a maintenance dose of 0.3-4mg/(kg*h). The infusion rate can be adjusted based on the sedation effect to achieve the appropriate level of sedation during EVT.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Patients receive perioperative sedation with dexmedetomidine
  Arms: the dexmedetomidine group
Drug: Midazolam — Patients receive perioperative sedation with midazolam
  Arms: the midazolam group

SUMMARY:
This study aims to conduct a multicenter, prospective, randomized clinical trial to scientifically evaluate the safety and efficacy of different perioperative sedation methods during endovascular thrombectomy in acute ischemic stroke patients with large vessel occlusion in the anterior circulation.

DETAILED DESCRIPTION:
In the perioperative period of endovascular thrombectomy, the main sedation options are midazolam (MDZ) and dexmedetomidine (DEX). Research has shown that both sedation methods have their advantages and disadvantages, and there is no consensus on how to choose between them. Therefore, this study aims to conduct a multicenter, prospective, randomized clinical trial to scientifically evaluate the safety and efficacy of different perioperative sedation methods during endovascular thrombectomy (EVT) in AIS patients with large vessel occlusion in the anterior circulation and hopes to contribute to the advancement of EVT in clinical practice.

In this trial, acute ischemic stroke patients with large vessel occlusion in the anterior circulation within 24 hours of symptom onset or last known well will be included. In the screening stage, participants who meet the inclusion criteria of the trial, upon completion of screening/baseline assessment and after signing the informed consent, will be randomly assigned in a 1:1 ratio to one of the following two treatment groups: the dexmedetomidine and midazolam conscious sedation groups. The primary end point is the proportion of modified Ranking score of 0-2 at 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Presenting with symptoms of acute ischemic stroke
3. CTA or MRA confirmed occlusion of the anterior circulation (intracranial carotid artery or M1, M2 segment of the middle cerebral artery)
4. Randomization finished within 24 hours of symptom onset or time last know well
5. Pre-stroke mRS score ≤2
6. NIHSS score ≥6 at the time of randomization
7. ASPECTS value ≥3
8. Informed consent signed

Exclusion Criteria:

General exclusion criteria

1. Pregnant or lactating women
2. Known allergy to contrast agents or nitinol devices
3. Known allergy to midazolam or other benzodiazepines
4. Known allergy to dexmedetomidine or its components
5. Planned to receive general anesthesia for EVT
6. Uncontrolled hypertension or hypotension (defined as systolic blood pressure >185 mmHg or < 90 mmHg, diastolic blood pressure >110 mmHg or < 60 mmHg)
7. Second-degree or third-degree heart blockage or bradyarrhythmia with a baseline heart rate lower than 50 beats/min
8. Any major surgery or serious trauma within 14 days
9. Known genetic or acquired bleeding diathesis (platelet count < 100\*109 /L, activated partial thromboplastin time > 50 s or international normalized ratio > 1.7)
10. Blood glucose <2.8 or > 22.2 mmol/L
11. Severe renal insufficiency (defined as glomerular filtration rate <30 ml/min or serum creatinine >220 mmol/L (2.5mg/dl))
12. Receiving hemodialysis or peritoneal dialysis
13. Life expectancy less than 1 year
14. Severe agitation or seizures
15. Clinical manifestations of central nervous system vasculitis
16. Premorbid neurological disease or mental disorders confounding evaluation
17. Unwilling to be followed up within 90 days
18. Participation in other interventional randomized clinical trials Imaging exclusion criteria

1. Evidence of intracranial hemorrhage on CT or MRI 2. Cerebellar infarction with obvious space-occupying effects and fourth ventricle compression on CT or MRI 3. Any untreated or incompletely treated intracranial aneurysm or any intracranial vascular malformation 4. Bilateral occlusion or multiple intracranial vessels occlusions 5. Intracranial tumors (with mass effect)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-06-13 (Estimated); Study Completion 2026-06-13 (Estimated)

PRIMARY OUTCOMES:
The proportion of mRS score 0-2 at 90 days | 90 days after randomization
  mRS is short for modified Ranking score (ranging from 0 to 6, with higher values indicating a worse functional outcome).

SECONDARY OUTCOMES:
Shift in the distribution of mRS scores at 90 days | 90 days after randomization
  mRS is short for modified Ranking score (ranging from 0 to 6, with higher values indicating a worse functional outcome).
The proportion of mRS score 0-1 at 90 days | 90 days after randomization
  mRS is short for modified Ranking score (ranging from 0 to 6, with higher values indicating a worse functional outcome).
The proportion of mRS score 0-3 at 90 days | 90 days after randomization
  mRS is short for modified Ranking score (ranging from 0 to 6, with higher values indicating a worse functional outcome).
Rates of successful recanalization | Immediately after the thrombectomy procedure is completed
  Successful recanalization is defined as mTICI≥2b. mTICI is short for modified Thrombolysis in cerebral Infarction (ranging from 0 to 3, with higher values indicating a better reperfusion state).
Score on the ASPECTS at 24-72 hours | 24-72 hours after randomization
  ASPECTS is short for Alberta Stroke Program Early CT Score (ranging from 0 to 10, with a higher score indicating a better perfusion state).
RASS score ≤ -3 during procedure | During operation
  Deep sedation defined as RASS score ≤ -3. RASS is short for Richmond Agitation and Sedation Scale. RASS is a score of the degree of sedation (range from -5 to +4, higher values indicate a worse sedation state).
RASS score ≤ 0 during procedure | During operation
  Under sedation defined as RASS score ≤ 0. RASS is short for Richmond Agitation and Sedation Scale. RASS is a score of the degree of sedation (range from -5 to +4, higher values indicate a worse sedation state).
Changes of the GCS score at 24 hours | 24 hours after randomization
  GCS is short for Glasgow Coma Scale. GCS is a score of the degree of comma (range from 3 to 15, higher values indicate more severe comma).
Changes of the NIHSS score at 24 hours | 24 hours after randomization
  NIHSS is short for National Institute of Health stroke scale. NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits).
Changes of the GCS score at 5-7 days | 5-7 days after randomization
  GCS is short for Glasgow Coma Scale. GCS is a score of the degree of comma (range from 3 to 15, higher values indicate more severe comma).
Changes of the NIHSS score at 5-7 days | 5-7 days after randomization
  NIHSS is short for National Institute of Health stroke scale. NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits).
Barthel Index at 90 days | 90 days after randomization
  Barthel Index is an ordinal disability score of 10 categories (range from 0 to 100, higher values indicate better prognosis)

OTHER OUTCOMES:
Rates of symptomatic intracranial hemorrhage at 48 hours | 48 hours after randomization
  Clinical safety endpoint. Intracranial hemorrhage within 48 hours on CT/MRI according to Heidelberg bleeding classification.
Rates of procedure-related complications | within 90 days from randomization
  Clinical safety endpoint
Rates of mortality at 90 days | within 90 days from randomization
  Clinical safety endpoint
Rates of adverse events | within 90 days from randomization
  Clinical safety endpoint
Rates of severe adverse events | with 90 days from randomization
  Clinical safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, Principal Investigator — Department of Neurology, Jinling Hospital, China
Locations (2):
- China (2):
  - Jinling Hospital, Medical School of Nanjing University, Nanjing, None Selected
  - The General Hospital of Western Theater Command PLA, Chengdu

IPD SHARING:
Plan to Share IPD: No